CLINICAL TRIAL: NCT02891200
Title: Comparing Effectiveness of Self-management and Peer Support Communication Programs Amongst Chronic Obstructive Pulmonary Disease (COPD) Patients and Their Family Caregivers
Brief Title: Impact of a Peer Support Program Amongst COPD Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00114571
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare professional (HCP) Arm (Experimental): Healthcare professional (HCP) Arm includes a trained respiratory therapist who will provide COPD self-management education and support via an in-person session and written materials .
  Interventions: Other: HCP support
- HCP plus Peer arm (Experimental): HCP plus Peer arm involves delivering of HCP support as in HCP Arm , along with adding Peer Support Program services. This program is offered to participants by especially trained 'peer mentors' with oversight from a social worker.
  Interventions: Other: Peer support program; Other: HCP support

INTERVENTIONS:
Other: Peer support program — The Peer Support Program offers education and support to participants by especially trained 'peer mentors' with oversight from a social worker.
  Arms: HCP plus Peer arm
Other: HCP support — Healthcare professional (HCP) support will be provided by a trained respiratory therapist who will provide COPD self-management education and support via an in-person session and written materials .

SUMMARY:
The study is to compare the effectiveness of two health communication and dissemination strategies that are designed to engage patients and family caregivers in successfully managing COPD in 'real-world' settings. Both strategies aim to advance patient understanding of COPD, its treatment options, and self-care tasks; support them in coping with the disease; and enable them to adopt a variety of positive behaviors, including adherence to treatment plans, smoking cessation, joining pulmonary rehabilitation programs, and assuming an active, healthy lifestyle. One strategy relies on the healthcare professional (HCP) as the primary communicator about COPD self-management (HCP arm), whereas the other uses a dual approach that involves both healthcare professionals and peer mentors delivering such communication (HCP plus Peer arm). Peer mentors are COPD patients and caregivers who have successfully managed COPD and have received foundational training on peer mentoring. Specifically, the study aims are to : 1) Conduct a randomized controlled trial in which the 'HCP' and 'HCP plus Peer' strategies are tested in 'real-world' healthcare settings; 2) compare the impact of these strategies on patient satisfaction, experience, activation, self- efficacy, self-care behavior, health status, quality of life, use of Emergency Department (ED) and hospital services, and survival; and, 3) compare the impact of these strategies on caregiver satisfaction, experience, self-efficacy, stress, and coping skills.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a prevalent global condition that results in high mortality, morbidity, symptom burden, and functional limitations that impact the quality of life. COPD is the third leading cause of death in the US and a leading cause of hospitalizations. COPD patients report unmet needs in regards to information about their disease and how to manage and cope with it at an intellectual, emotional, and social level. Many COPD patients lack the information and skills that they need to correctly use their inhaled medications, manage 'breathlessness episodes', and detect early signs of a COPD exacerbation. Pulmonary rehabilitation programs are established to help COPD patients increase their exercise capacity and reduce fatigue and dyspnea with daily activity. While clinical trials testing these programs have demonstrated significant improvements in health-related quality of life and reduced dyspnea and fatigue amongst participants, it remains unclear how best to engage and motivate patients to participate in them.

Self-management support interventions which involve "collaboratively helping patients acquire and practice the skills needed to carry out disease-specific medical regimens, change their health behavior to adjust their roles for optimal function, improve day-to-day control of their disease, and improve their well-being", have been demonstrated in several trials to improve health-related quality of life, and reduce symptom burden, hospitalizations, and ED visits amongst COPD patients. However, it is still unclear which self-management support strategies employed in 'real world' settings are most effective in engaging, motivating, and enabling patients to successfully follow recommended treatments, adopt desired health behaviors, and thus achieve the desired improvements in their health outcomes.

The planned study design is a single- blinded randomized controlled trial to compare the effectiveness of two strategies for engaging and supporting COPD patients and their family caregivers in self-management of COPD. The two strategies/study arms are: 1) the 'HCP arm' where the healthcare professional (HCP) is the primary communicator about COPD self-management with the patient participants; and 2) the 'HCP plus Peer arm', where both healthcare professionals and peer mentors engage with study participants in conversations about COPD self-management using multiple channels including one- to- one and group conversations. Participants will be randomized in a 1:1 ratio into the two study arms. The trial will be conducted amongst COPD patients coming to the hospital or clinic at two study sites within Johns Hopkins Healthcare System. Recruitment from both sites and multiple settings allows for a more representative COPD patient population to be enrolled in the study, thus increasing the external validity of study findings.

The research study will answer the research question: Amongst COPD patients and their caregivers, would a dual strategy that combines healthcare professional and peer mentor delivery of COPD self- management education and support result in greater improvements in health status and quality of life, and reductions in acute healthcare services' utilization, compared to relying on healthcare professionals alone in these communications? Would such dual strategy result in reduced caregiver stress and improved coping and satisfaction? The study hypothesis is that the dual strategy of using 'HCP plus peer support' to engage and support COPD patients and caregivers will have superior outcomes to the 'HCP only' strategy in the following areas : a) Improved health- related quality of life and reduced numbers of COPD-related hospital and ED visits; b) improved patient activation, self-efficacy, and self-care behaviors; c) improved family caregivers' satisfaction and self- efficacy. These improvements will be noted at 3, 6, and 9 months compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Has a physician diagnosis of COPD AND is on treatment for it ( defined as receiving treatment at hospital or clinic for COPD)

Exclusion Criteria:

* Cognitive dysfunction impairing ability to provide informed consent and follow instructions
* Active substance abuse or unstable psychiatric condition
* Terminal illness (i.e. less than 6 months life expectancy) that is non-COPD related
* Planning to move from area
* Living at a facility, such as Hospice or nursing home
* Unable to provide contact information
* Does not understand English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Aboumatar, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aboumatar H, Garcia Morales EE, Jager LR, Naqibuddin M, Kim S, Saunders J, Bone L, Linnell J, McBurney M, Neiman J, Riley M, Robinson N, Rand C, Wise R. Comparing Self-Management Programs with and without Peer Support among Patients with Chronic Obstructive Pulmonary Disease: A Clinical Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1687-1696. doi: 10.1513/AnnalsATS.202108-932OC. PMID 35442179

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthcare Professional (HCP) Arm: Healthcare professional (HCP) Arm includes a trained respiratory therapist who will provide Chronic Obstructive Pulmonary Disease (COPD) self-management education and support via an in-person session and written materials .
  HCP support: Healthcare professional (HCP) support will be provided by a trained respiratory therapist who will provide COPD self-management education and support via an in-person session and written materials .
Period: Overall Study
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Started | 145 | 147
Completed | 103 | 98
Not Completed | 42 | 49
Not completed — Lost to Follow-up | 31 | 36
Not completed — Death | 10 | 9
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm | Total
Number analyzed (Participants) | 145 | 147 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.5) | 67.5 (9.3) | 67.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 85 | 179
  Male | 51 | 62 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 34 | 76
  White | 101 | 106 | 207
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Total Score for St. George Respiratory Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured using the St. George Respiratory Questionnaire. Score ranges from 0 to 100. Higher score indicates a worse quality of life.
  units on a scale | 55.0 (20.0) | 56.3 (18.0) | 55.6 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Health-related Quality of Life at 6 Months
Description: Change in health-related quality of life (HRQoL) at 6 months post-enrollment from baseline. The HRQoL is measured using the St. George Respiratory Questionnaire (SGRQ), a validated instrument that will be administered to participant by a trained research team member. SGRQ measures health-related quality of life among patients with respiratory diseases. It is a 40 items questionnaire grouped into three domains (Symptoms, Activity, and Impacts). The overall summary score is calculated by summing the weights of all items with positive response in the questionnaire and dividing that by sum of weights for all items, times 100. Total scores range from 0 to 100. Higher score reflect worse quality of life and a decrease in score indicates improvement HRQoL . Change in score was calculated as the total score at 6 month post-enrollment minus total score at baseline ( i.e at enrollment ). Minimum clinically important difference (MCID) for SGRQ is a 4-point improvement (i.e decrease in score).
Time Frame: enrollment to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 144 | 143
units on a scale | -1.78 (19.7) | -0.52 (18.3)
Statistical Analysis 1: Comparison: Healthcare Professional (HCP) Arm vs HCP Plus Peer Arm; Test type: Superiority; p = 0.467, Mixed Models Analysis; Mixed effects linear model with study site and setting as fixed effects, and adjusted for baseline SGRQ domain scores; Predicted Mean Difference = 1.46, 95% CI 2-sided [-2.47 to 5.38]

2. Secondary Outcome: Combined Number of COPD-related Hospitalizations and ED Visits Per Participant at 6 Months
Description: All hospitalizations and ED visits discharge diagnoses are reviewed and those that are COPD-related are counted from time of participant enrollment into study till 6 months afterwards. A visit is coded as COPD-related if:
  1. The principle discharge diagnosis was any of the following : J41.0 ; J41.1; J41.8; J42; J43.0; J43.1; J43.2; J43.8; J43.9; J44.0; J44.1; J44.9.
     Or
  2. The principle discharge diagnosis was respiratory failure AND the visit had a secondary diagnosis of J44.0 or J44.1 . The respiratory failure codes are J96.00; J96.01; J96.02; J96.20; J96.21; J96.22; J96.90; J96.91; J96.92; R06.03; R09.2 .
Time Frame: Measured at 6 months post enrollment
Population: Patients who have passed away or withdrew before 6 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: COPD-related visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 135 | 137
COPD-related visits per participant | 0.79 [0.30 to 1.2] | 0.62 [0.34 to 0.9]

3. Secondary Outcome: Combined Number of COPD-related Hospitalizations and ED Visits Per Participant at 9 Months
Description: All hospitalizations and ED visits discharge diagnoses are reviewed and those that are COPD-related are counted from time of participant enrollment into study till 9 months afterwards. A visit is coded as COPD-related if:
  1. The principle discharge diagnosis was any of the following : J41.0 ; J41.1; J41.8; J42; J43.0; J43.1; J43.2; J43.8; J43.9; J44.0; J44.1; J44.9.
     Or
  2. The principle discharge diagnosis was respiratory failure AND the visit had a secondary diagnosis of J44.0 or J44.1 . The respiratory failure codes are J96.00; J96.01; J96.02; J96.20; J96.21; J96.22; J96.90; J96.91; J96.92; R06.03; R09.2 .
Time Frame: Measured at 9 months post enrollment
Population: Patients who have passed away or withdrew before 9 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: COPD-related visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 120 | 130
COPD-related visits per participant | 1.06 [0.22 to 1.9] | 1.02 [0.45 to 1.6]

4. Secondary Outcome: Combined Number of COPD-related Hospitalizations and ED Visits Per Participant at 3 Months
Description: All hospitalizations and ED visits discharge diagnoses are reviewed and those that are COPD-related are counted from time of participant enrollment into study till 3 months afterwards. A visit is coded as COPD-related if:
  1. The principle discharge diagnosis was any of the following : J41.0 ; J41.1; J41.8; J42; J43.0; J43.1; J43.2; J43.8; J43.9; J44.0; J44.1; J44.9.
     Or
  2. The principle discharge diagnosis was respiratory failure AND the visit had a secondary diagnosis of J44.0 or J44.1 . The respiratory failure codes are J96.00; J96.01; J96.02; J96.20; J96.21; J96.22; J96.90; J96.91; J96.92; R06.03; R09.2 .
Time Frame: Measured at 3 months post enrollment
Population: Patients who have passed away or withdrew before 3 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: COPD-related visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 140 | 142
COPD-related visits per participant | 0.41 [0.16 to 0.6] | 0.27 [0.15 to 0.3]

5. Secondary Outcome: Combined Number of All-cause Hospitalizations and ED Visits Per Participant at 6 Months
Description: All hospitalizations and ED visits will be counted from time of participant enrollment into study till 6 months afterwards.
Time Frame: Measured at 6 months post enrollment
Population: Patients who have passed away or withdrew before 6 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 135 | 137
visits per participant | 1.32 [0.52 to 2.1] | 1.07 [0.58 to 1.5]

6. Secondary Outcome: Combined Number of All-cause Hospitalizations and ED Visits Per Participant at 9 Months
Description: All hospitalizations and ED visits will be counted from time of participant enrollment into study till 9 months afterwards.
Time Frame: Measured at 9 months post enrollment
Population: Patients who have passed away or withdrew before 9 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 120 | 130
visits per participant | 1.79 [0.47 to 3.1] | 1.65 [0.82 to 2.4]

7. Secondary Outcome: Combined Number of All-cause Hospitalizations and ED Visits Per Participant at 3 Months
Description: All hospitalizations and ED visits will be counted from time of participant enrollment into study till 3 months afterwards.
Time Frame: Measured at 3 months post enrollment
Population: Patients who have passed away or withdrew before 3 months from enrollment are excluded from the analysis
Measure: Mean (95% Confidence Interval); unit: visits per participant
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 140 | 142
visits per participant | 0.71 [0.3 to 1.11] | 0.53 [0.3 to 0.76]

8. Secondary Outcome: Change in Health-related Quality of Life at 9 Months
Description: Change in health-related quality of life (HRQoL) at 9 months post-enrollment from baseline. The HRQoL is measured using the St. George Respiratory Questionnaire (SGRQ), a validated instrument that will be administered to participant by a trained research team member. SGRQ measures health-related quality of life among patients with respiratory diseases. It is a 40 items questionnaire grouped into three domains (Symptoms, Activity, and Impacts). The overall summary score is calculated by summing the weights of all items with positive response in the questionnaire and dividing that by sum of weights for all items, times 100. Total scores range from 0 to 100. Higher score reflect worse quality of life and a decrease in score indicates improvement HRQoL . Change in score was calculated as the total score at 9 month post-enrollment minus total score at baseline ( i.e at enrollment ). Minimum clinically important difference (MCID) for SGRQ is a 4-point improvement (i.e decrease in score).
Time Frame: enrollment to 9 months
Population: The Number of Participants Analyzed for change in quality of life at 9 months is different from that at 6 months because not all participants were candidates to receive the 9 months quality of life measurement due to end of project period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 144 | 143
units on a scale | 2.27 (23.29) | 4.61 (20.83)

9. Secondary Outcome: Mortality Rate
Description: Assessed at 6 months
Time Frame: Measured at 6 months post enrollment
Population: Patients who withdrew from study are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 144 | 143
Participants | 10 | 9

10. Secondary Outcome: Mortality Rate
Description: Assessed at 9 months
Time Frame: Measured at 9 months post enrollment
Population: Patients who withdrew from study are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 144 | 143
Participants | 15 | 13

11. Secondary Outcome: Mortality Rate
Description: Assessed at 3 months
Time Frame: Measured at 3 months post enrollment
Population: Patients who withdrew from study are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
Number analyzed (Participants) | 144 | 143
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: 9 months post enrollment
Description: Deaths were systematically assessed. Serious adverse events were assessed systematically for all hospitalizations. Other serious adverse events were tracked based on reports by patient or study interventionists. Reported adverse events results are for all participants except those who withdrew from study (total of 5). Reasons for withdrawal included administrative dis-enrollment (n=2) and patient desire due to reported data collection burden (n=3).
Arm/Group | Healthcare Professional (HCP) Arm | HCP Plus Peer Arm
All-Cause Mortality (participants affected / at risk) | 15/144 | 13/143
Serious Adverse Events (participants affected / at risk) | 57/144 | 57/143
Other Adverse Events (participants affected / at risk) | 0/144 | 0/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthcare Professional (HCP) Arm (N=144) | HCP Plus Peer Arm (N=143)
Hospitalizations for any cause (General disorders) | 57 | 57 — These events are hospitalizations of any cause that occurred during the study period (between study enrollment and 9 months). These are anticipated adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT02891200/Prot_SAP_000.pdf